CLINICAL TRIAL: NCT03865693
Title: Effects of Pain Scrambler Therapy for the Alterations of Cerebral Blood Volume in Pain Network of Neuropathic Pain on Burn Patients
Brief Title: Effects of Pain Scrambler Therapy for the Alterations of Cerebral Blood
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hangang Sacred Heart Hospital (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HangangSHH-3
Record Dates: First submitted 2019-03-05; First posted 2019-03-07 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Pain, Neuropathic
Keywords: Burn; pain scrambler
MeSH Terms: conditions — Neuralgia; Burns

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- scarmbler treatment group (Experimental): Each Scrambler therapy with the MC5-A Calmare® therapy device (Competitive Technologies, Inc. Fairfield, USA ) was performed for 40 min daily (Monday through Friday) for 10 consecutive days. The experimental participants were received scarmbler therapy 10 times for 2 weeks. The stimulus was increased to the maximum intensity bearable by the individual patient without causing any additional pain or discomfort.
  Interventions: Device: scarmbler therapy
- sham treatment group (Sham Comparator): conservative management without scarmbler therapy
  Interventions: Device: scarmbler therapy

INTERVENTIONS:
Device: scarmbler therapy — Scrambler therapy is a patient-specific electrocutaneous nerve stimulation device.

SUMMARY:
Prevalence of chronic pain has been shown to be high after thermal injury. Post-burn neuropathic pain causes chronic disabilities that is often difficult to treat effectively. Pain Scrambler therapy is a patient-specific electrocutaneous nerve stimulation device. To study changes in the pain network associated with neuropathic pain, magnetic resonance imaging(MRI) was used to evaluate cerebral blood volume(CBV) in patients who had been injuried by burn. Participants (N=40, experimental 20 and control group 20) comprised patients with neuropathic pain after thermal injury. The subjects complained of severe neuropathic pain that was rated at least 5 on the visual analogue scale (VAS), despite treatments with gabapentin medication and other physical modalities. Each Scrambler therapy with the MC5-A Calmare® therapy device (Competitive Technologies, Inc. Fairfield, USA ) was performed for 40 min daily (Monday through Friday) for 10 consecutive days. The stimulus was increased to the maximum intensity bearable by the individual patient without causing any additional pain or discomfort. The intensity of neuropathic pain was measured using the visual analogue scale(VAS). Depressive mood was assessed using the Beck Depression Scale. Voxel-wise comparisons of relative CBV maps were made between before scrambler therapy and after 10 scrambler therapy sessions over the entire brain volume. The relationship between individual participant CBV(measured in voxels), BDS and VAS score was also examined. We observed decreased in the cerebral pain network of patients with burn injury. Scrambler therapy is a non-invasive, non-medicinal modality that significantly reduced burn-associated neuropathic pain. Scrambler therapy should be considered as a treatment option for burn survivors with severe neuropathic pain.

DETAILED DESCRIPTION:
The groups (scrambler therapy and sham therapy) were randomly assigned. All subjects were recruited in scrambler thrapy and sham stimulation. Main study outcomes included group differences in CBV changed and the the relationship between CBV changes and neuropathic pain intensity. These analyses were performed using the same framework of the general linear model, which was repeatedly applied to each voxel with the same coordinates.

ELIGIBILITY:
Inclusion Criteria:

* Burn patients
* severe neuropatic pain rated at least 5 on the 10-point numerical rating scale (NRS)

Exclusion Criteria:

* cardiac arrest history
* history of neurologi disease or brain surgery
* unstable heart disease or presence of a cardiac pacemaker
* pain resulting from other causes like as neuromuscular diseases
* psychiatric disorder
* diabetes mellitus
* abnormal renal function
* contraindication for MRI, or pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
neuropathic pain score | after 4 weeks scrambler therapy
  visual analog scale, Zero ("0") represented no pain and 10 represented unbearable symptoms

SECONDARY OUTCOMES:
Cerebral blood volume | after 4 weeks scrambler therapy
  Cerebral blood volume(CBV) is a hemodynamic variable that is highly correlated with oxygen metabolism, representing the fraction of cerebral tissue volume occupied by blood at a given time point.

CONTACTS AND LOCATIONS:
Overall Officials: Cheong Hoon Seo, M.D., Principal Investigator — Hangang Sacred Heart Hospital
Locations (1):
- Hangang Sacred Heart Hospital, Seoul, Yeong-deungpo-Dong, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
after review

REFERENCES:
- [Background] Joo SY, Cho YS, Cho SR, Kym D, Seo CH. Effects of pain Scrambler therapy for management of burn scar pruritus: A pilot study. Burns. 2017 May;43(3):514-519. doi: 10.1016/j.burns.2016.09.028. Epub 2016 Oct 15. PMID 27756587
- [Result] Majithia N, Smith TJ, Coyne PJ, Abdi S, Pachman DR, Lachance D, Shelerud R, Cheville A, Basford JR, Farley D, O'Neill C, Ruddy KJ, Sparadeo F, Beutler A, Loprinzi CL. Scrambler Therapy for the management of chronic pain. Support Care Cancer. 2016 Jun;24(6):2807-14. doi: 10.1007/s00520-016-3177-3. Epub 2016 Apr 4. PMID 27041741
- [Derived] Lee SY, Park CH, Cho YS, Kim L, Yoo JW, Joo SY, Seo CH. Scrambler Therapy for Chronic Pain after Burns and Its Effect on the Cerebral Pain Network: A Prospective, Double-Blinded, Randomized Controlled Trial. J Clin Med. 2022 Jul 22;11(15):4255. doi: 10.3390/jcm11154255. PMID 35893347